CLINICAL TRIAL: NCT06263582
Title: Pharmacokinetics of Intravaginal, Self-administered Artesunate Vaginal Pessaries Among Women in Kenya
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGHID12333; K12HD103085 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Cervix Cancer; Cervix Intraepithelial Neoplasia Grade 3; Cervix; Intraepithelial Neoplasia, Grade I; Cervix; Intraepithelial Neoplasia, Grade II
Keywords: Artesunate; dihydroartemisinin; pharmacokinetics
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Carcinoma in Situ; Lymphoma, Follicular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artesunate vaginal inserts/ pessaries (Experimental): Artesunate vaginal inserts/pessaries are used as a treatment for cervical precancerous lesions.
  Interventions: Drug: Artesunate pessary; Diagnostic Test: blood draws for pharmacokinetics of the study drug

INTERVENTIONS:
Drug: Artesunate pessary — Subjects will use the study pessaries, placed in the vagina every day for 5 consecutive days.
Diagnostic Test: blood draws for pharmacokinetics of the study drug — On day 5, all participants will have their blood draws before they use the pessary, and at 15 min, 30 mins, 1 hour, 2 hours, 4 hours, 6 hours, and 8 hours after inserting the pessary. Blood samples will be tested for the pharmacokinetics of the study drug.

SUMMARY:
This study investigates the pharmacokinetics of Artesunate (AS) and dihydroartemisinin (DHA), the active metabolite of Artesunate, following intravaginal use at the dosing and frequency being studied for cervical precancer treatment. A secondary objective is to investigate safety among study participants.

DETAILED DESCRIPTION:
Due to lack of access to primary and secondary prevention, women living in low-and middle-income countries bear a disproportionate burden of cervical cancer, accounting for 90% of new cases and 85% of deaths globally. Cervical cancer can be prevented through vaccination against Human papillomavirus (HPV), whose infection is required to develop cervical cancer. Among unvaccinated women, screening for HPV or cervical precancer allows identification of precancerous lesions - primarily cervical intraepithelial neoplasia grade 2 or 3 (CIN2/3), that can be treated and cured, to prevent progression to cancer. Most CIN2/3 lesions that are left untreated will progress to invasive cervical cancer. Current treatments for CIN2/3 in both high- and low-resource countries (LMICs) require trained health care providers, who are often out of reach for many women, particularly in rural areas in LMICs. Lack of access to precancer treatment following screening in LMICs in part accounts for the high burden of incident cervical cancer. Preclinical data have demonstrated pro-apoptotic effects of Artesunate (AS), a commonly available drug with an excellent safety profile in oral, rectal and intravenous routes primarily used to treat malaria in LMICs. This led to a recent Phase I study in the United States that demonstrated that self-administered vaginal artesunate inserts (pessaries) are safe, well-tolerated, and demonstrate efficacy for treatment of CIN2/3. Based on the mechanism of action, the clinical safety profile, and widespread availability as a generic drug on the World Health Organization (WHO) List of Essential Medications, vaginal artesunate inserts (pessaries), if backed by data from randomized trials, may offer patient-controlled and access cervical precancer treatment method for women in LMICs who face the greatest burden of cervical cancer and have difficulty accessing skilled providers for precancer treatment. However, given that artesunate is a well-known drug used in malaria treatment, it is critical to ensure that vaginal application of the drug will not promote resistance for use in malaria treatment.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older
2. Negative pregnancy test at screening
3. Willingness to use contraception (hormonal or barrier) during the 5-day study dosing phase if of childbearing age (less than 50 years of age)
4. Ability and willingness to provide informed consent.

Exclusion Criteria

1. Current pregnancy or breastfeeding status
2. History of total hysterectomy
3. Known allergy to Artesunate.
4. Have a medical comorbidity that in the opinion of the investigator would interfere with study participation.
5. Currently receiving artemisinin-based agents for malaria treatment or completed artemisinin-based treatment within the previous 3 days.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are eligible
Enrollment: 12 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chemtai Mungo, MD, MPH, FACOG, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lumumba Sub-County Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in one center in Kenya.
Pre-assignment Details: Twelve participants consented and found eligible.
Period: Overall Study
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 12
Level of education [Count of Participants; unit: Participants]
  College or higher | 2
  Completed Secondary | 10
Occupation [Count of Participants; unit: Participants]
  Salaried work | 1
  other | 1
  student | 10
Marital Status [Count of Participants; unit: Participants]
  Single/Never Married | 12
  Married | 0
Electricity available [Count of Participants; unit: Participants]
  yes | 11
  no | 1
Tap water available [Count of Participants; unit: Participants]
  yes | 10
  No | 2
Current or prior tobacco use [Count of Participants; unit: Participants]
  yes | 2
  No | 10
Current or prior alcohol use [Count of Participants; unit: Participants]
  Yes | 9
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Area Under the Plasma Concentration Versus Time Curve (AUC) of Dihydroartemisinin
Description: To determine the area under the plasma concentration versus time curve (AUC) of dihydroartemisinin (DHA) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries). Mean DHA AUC will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/mL-h
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
ng/mL-h | 464.90 (228.70)

2. Secondary Outcome: To Determine the Area Under the Plasma Concentration Versus Time Curve (AUC) of Artesunate (AS)
Description: To determine the area under the plasma concentration versus time curve (AUC) of Artesunate (AS) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries). Mean artesunate AUC will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/mL-h
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
ng/mL-h | 504.21 (281.11)

3. Secondary Outcome: To Determine the Maximum Concentration of Artesunate (AS)
Description: To determine the maximum concentration of Artesunate (AS) (Cmax) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean artesunate Cmax (ng/ml) value will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
ng/mL | 83.74 (42.73)

4. Secondary Outcome: To Determine the Maximum Concentration of Dihydroartemisinin (DHA) (Cmax)
Description: To determine the maximum concentration of dihydroartemisinin (DHA) (Cmax) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean DHA Cmax (ng/ml) value will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
ng/mL | 97.00 (53.12)

5. Secondary Outcome: To Determine the Time to Maximum Concentration (Tmax) of Artesunate (AS) Following Five Consecutive Days
Description: To determine the time to maximum concentration (Tmax) of Artesunate (AS) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean DHA Tmax (hours) value will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
hours | 4.17 (1.59)

6. Secondary Outcome: To Determine the Time to Maximum Concentration (Tmax) of Dihydroartemisinin (DHA
Description: To determine the time to maximum concentration (Tmax) of dihydroartemisinin (DHA) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean (Tmax) will be submitted.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
hours | 6.33 (1.67)

7. Secondary Outcome: To Determine the Half-life (t1/2) of Artesunate (AS)
Description: To determine the half-life (t1/2) of Artesunate (AS) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women. Mean Artesunate half-life (t1/2) (mins) will be submitted.
Time Frame: Day 5
Population: The plasma half-life of Artesunate could not be estimated because the concentration versus time profiles did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration of intravaginal artesunate.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

8. Secondary Outcome: To Determine the Half-life (t1/2) of Dihydroartemisinin (DHA)
Description: To determine the half-life (t1/2) of dihydroartemisinin (DHA) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean DHA half-life (mins) will be submitted.
Time Frame: Day 5
Population: The plasma half-life of dihydroartemisinin (DHA) could not be estimated because the concentration versus time profiles did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

9. Secondary Outcome: To Determine the Apparent Clearance (CL/F) of Artesunate (AS)
Description: To determine the apparent clearance (CL/F) of Artesunate (AS) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean Artesunate clearance (L/Kg/hr) will be submitted.
Time Frame: Day 5
Population: The plasma apparent clearance (CL/F) of Artesunate could not be estimated because the concentration versus time profiles of both forms did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration of intravaginal artesunate.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

10. Secondary Outcome: To Determine the Apparent Clearance (CL/F) of Dihydroartemisinin (DHA)
Description: To determine the apparent clearance (CL/F) of dihydroartemisinin (DHA) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean DHA clearance (L/Kg/hr) will be submitted.
Time Frame: Day 5
Population: The plasma apparent clearance (CL/F) of dihydroartemisinin (DHA) could not be estimated because the concentration versus time profiles of both forms did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

11. Secondary Outcome: To Determine the Volume of Distribution (V/F) of Artesunate (AS)
Description: To determine the volume of distribution (V/F) of Artesunate (AS) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean Artesunate volume of distribution (L/Kg) will be submitted.
Time Frame: Day 5
Population: The plasma volume of distribution (V/F) of Artesunate (AS) could not be estimated because the concentration versus time profiles of both forms did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration of intravaginal artesunate.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

12. Secondary Outcome: To Determine the Volume of Distribution (V/F) of Dihydroartemisinin (DHA)
Description: To determine the volume of distribution (V/F) of dihydroartemisinin (DHA) following five consecutive days of self-administration of 200mg Artesunate vaginal inserts (pessaries) among healthy women.
  Mean dihydroartemisinin (DHA) of distribution (V/F) will be submitted.
Time Frame: Day 5
Population: The plasma volume of distribution (V/F) of dihydroartemisinin (DHA) could not be estimated because the concentration versus time profiles of both forms did not reach an elimination phase (i.e., the concentration versus time profile did not decrease) from 0 to 8h post administration.
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 0

13. Secondary Outcome: Type, Frequency, Severity, and Duration of Adverse Events
Description: To investigate the safety of a 5-day course of self-administered intravaginal artesunate vaginal inserts (pessary) in women. Type, frequency, severity, and duration of reported and observed adverse events (AEs) using the U.S National Cancer Institute Common Terminology Criteria for Adverse Events, v5.0 (CTCAE 5.0) and the Division of AIDS Female Genital Adverse Events Grading Table will be submitted.
Time Frame: Up to day 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
Number analyzed (Participants) | 12
Participants
  abdominal pain Grade 1 | 3
  vaginal discharge Grade 1 | 8
  Toothache- Grade 1 | 1
  vaginal fistula- Grade 2 | 1
  vaginal pruritis- Grade 1 | 1

ADVERSE EVENTS:
Time Frame: Up to ten days after the study intervention (vaginal insertion of Artesunate pessaries).
Description: AEs were collected according to National Cancer Institute Common Terminology Criteria for Adverse Events, v5.0 (CTCAE 5.0)
Arm/Group | Artesunate Vaginal Inserts/ Pessaries
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artesunate Vaginal Inserts/ Pessaries (N=12)
Abdominal Pain (Gastrointestinal disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 8
Toothache (Gastrointestinal disorders) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Pain in the extremity (Musculoskeletal and connective tissue disorders) | 1
Vaginal pruritis (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
Pharmacokinetic (PK) sampling from 0 to 8 hours after intravaginal administration of artesunate was not sufficient to capture the elimination phase of the drug and its metabolite. As a result, key plasma pharmacokinetic parameters including apparent clearance (CL/F), apparent volume of distribution (Vd/F), elimination half-life (t½), and area under the concentration-time curve from time zero to infinity (AUC₀-∞) could not be estimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT06263582/Prot_SAP_000.pdf